CLINICAL TRIAL: NCT05846113
Title: Renasight Clinical Application, Review and Evaluation (RenaCARE) Study
Acronym: RenaCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-048-TRP
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Kidney Diseases
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renacare patients (Experimental): Male or female patients, age 18 years or older at the time of signing the informed consent form (ICF). If over the age of 65, patient must have a family history of CKD or clinical suspicion of genetic disorder.
  Diagnosis of kidney disease
  Interventions: Diagnostic Test: Renasight

INTERVENTIONS:
Diagnostic Test: Renasight — The Renasight™ test is a next generation sequencing (NGS) gene mutation assay for patients with chronic kidney disease (CKD) which utilizes genomic DNA from patient blood or buccal swab samples to analyze over 380 genes that are associated with autosomal dominant, autosomal recessive and X-linked disorders.
  Patients undergoing Renasight™ testing are offered optional genetic information sessions in addition to their test results.
  RenasightTM is a commercially available Laboratory Developed Test (LDT) certified under the Clinical Laboratory Improvement Amendments (CLIA). This test has not been cleared or approved by the U.S. Food and Drug Administration (FDA).

SUMMARY:
This study is an open-label, multi-center study evaluating the clinical utility of Renasight in the diagnosis and management of kidney disease.

DETAILED DESCRIPTION:
Patients who are prospectively enrolled in the study will have blood or buccal swab samples sent to the Natera clinical lab for Renasight testing at the time of enrollment. Physicians will receive Renasight test results which may be used in clinical decision-making. At enrollment and at 1 month and 1 year following enrollment, clinical data will be submitted, and physician and subject questionnaires will be completed. Additional clinical follow-up and patient questionnaires may be completed at 2 and 3 years following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following selection criteria to be eligible for the study. Eligibility will be assessed by the investigator:

  1. Male or female patients, age 18 years or older at the time of signing the informed consent form (ICF). If over the age of 65, patient must have a family history of CKD or clinical suspicion of genetic disorder.
  2. Able to read, understand, and provide written informed consent
  3. Willing and able to comply with the study-related procedures
  4. Diagnosis of kidney disease, and/or one of the following without any kidney biopsy (note: can be newly diagnosed or existing patient):

     1. Nephropathy associated with Diabetes Mellitus (DM)*
     2. Nephropathy associated with Hypertension*
     3. Cystic nephropathy*
     4. Congenital nephropathy
     5. Tubulointerstitial disease of unknown etiology
     6. Proteinuric disease suggestive of a primary glomerulopathy by clinical evaluation
     7. Early, severe or familial hypertension
     8. Thrombotic microangiopathy
     9. Electrolyte and acid base disorder
     10. Nephrolithiasis with family history
     11. CKD of unknown cause after standard nephrological evaluation
     12. End stage kidney disease (ESRD) *Total number of patients in each of these categories will not exceed 10% of total cohort

Exclusion Criteria:

* Patients are not eligible for the study if they meet any of the following criteria, as assessed by the investigator:

  1. Age less than 18, or greater than 65 without a family history of CKD or clinical suspicion of genetic disorder
  2. History of renal transplant
  3. Clinical features and a kidney biopsy diagnosis strongly indicative of a secondary nephropathy (e.g., diabetic nephropathy, lupus nephritis, acute kidney injury)
  4. Previously confirmed diagnosis of a hereditary kidney disease via genetic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1720 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Test Positive Prevalence: The frequency of positive test results across the entire cohort and within different categories of kidney disorders will be analyzed. | Within 3 months of recruitment close
  Frequency of positive test results is defined as the number of patients in a given category with a genetic finding on Renasight divided by the total number of patients in that category. Changes in diagnosis from baseline physician questionnaire to post-result physician questionnaire will be classified
Frequency of positive test results of Renasight compared to frequency of positive test results of phenotypic panels | Within 6 months of recruitment close
  The frequency of positive test results of the Renasight panel will be compared to phenotype-specific commercial panels virtually reconstructed from the Renasight gene content. The frequency of positive test results will also be compared across different clinical categories of disease in the study population.
Number of participants with changed treatment or clinical management and new clinical diagnoses established based on Renasight test results. | Within 3 years and 6 months of recruitment close
  The enrolling physician will complete baseline questionnaires, 1-month post-result questionnaires, and 1-year follow-up questionnaires. Changes to pre-result planned management as well as new diagnostic information will be assessed. Pre-result and post-result surveys will be reviewed for all subjects, regardless of test results.

SECONDARY OUTCOMES:
Evaluate the impact of Renasight on patient satisfaction, health knowledge and genetics literacy. | Within 2 years of recruitment close
  Pre- and post-results questionnaires will be assessed for associations between genetic testing and psychological wellbeing and the impact on genetic testing on healthcare utilization. Genetic literacy pre- and post-results will be compared.
Evaluate the impact of Renasight on family outcomes. | Within 2 years of recruitment close
  Results of the post-results survey will be analyzed to determine the number of family members who have undergone screening and diagnosis as a result of genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Hoss Tabriziani, MD, Principal Investigator — Natera, Inc.
Locations (31):
- United States (31):
  - Liberty Dialysis/US Renal Care (USRC), Anchorage, Alaska
  - AKDHC Medical Research Services, LLC (Arizona Kidney Disease & Hypertension Centers), Tucson, Arizona
  - Renal Consultants Medical Group (USRC), Granada Hills, California
  - California Institute of Renal Research (CIRR)/(Balboa), San Diego, California
  - Western Nephrology and Metabolic Bone Disease, PC, Arvada, Colorado
  - Yale University, New Haven, Connecticut
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Nephrology & Hypertension Specialists, PC (USRC), Dalton, Georgia
  - Nephrology Associates of Northern Illinois (NANI), Hinsdale, Illinois
  - Nephrology Associates of Northern Indiana (NANI), Fort Wayne, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - USRC Kidney Research (USRC), Gallup, New Mexico
  - NYU Langone Hospital-Long Island, Mineola, New York
  - PRINE Health, New Hyde Park, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - Renal Care Consultants, P.C., Johnstown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - US Renal Care (USRC), San Antonio, Texas
  - Kidney & Hypertension Transplant Associates, San Antonio, Texas
  - Texas Kidney Care, San Antonio, Texas
  - South Texas Renal Care Group (USRC), San Antonio, Texas
  - US Renal Care (USRC) - Westover Hills, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chebib FT, Wang X, Udani SM, Westemeyer M, Clark D, Zhang Z, Bloom MS, Milo Rasouly H, Kolupaeva V, Mizani MR, Dossabhoy NR, Faravardeh A, Demko ZP, Kotte S, Punj S, Chapman SL, Rabinowitz M, Schneider R, Tabriziani H, Bhorade S, Gharavi AG, Dahl NK. Genetic Testing in the Management of Adult CKD. J Am Soc Nephrol. 2025 Oct 29. doi: 10.1681/ASN.0000000913. Online ahead of print. No abstract available. PMID 41563380
- [Derived] Dahl NK, Bloom MS, Chebib FT, Clark D, Westemeyer M, Jandeska S, Zhang Z, Milo-Rasouly H, Kolupaeva V, Marasa M, Broumand V, Fatica RA, Raj DS, Demko ZP, Marshall K, Punj S, Tabriziani H, Bhorade S, Gharavi AG. The Clinical Utility of Genetic Testing in the Diagnosis and Management of Adults with Chronic Kidney Disease. J Am Soc Nephrol. 2023 Dec 1;34(12):2039-2050. doi: 10.1681/ASN.0000000000000249. Epub 2023 Oct 5. PMID 37794564